CLINICAL TRIAL: NCT03185260
Title: International Registry of Laypeople's CPR Performance After Training With Feedback Devices
Brief Title: Registry of Laypeople's CPR Performance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pavia nel Cuore (Other)
Collaborators: Robbio nel Cuore (Unknown)
Responsible Party: Principal Investigator, Enrico Baldi, President, M.D., Pavia nel Cuore
Other Study IDs: FeedbackRegistry
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Quality of Cardio-pulmonary Resuscitation
Keywords: Cardio-Pulmonary Resuscitation; Cardiac Arrest; Training
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the registry is to collect laypeople's performance after a BLS/AED course carried out with the use of feedback devices.

DETAILED DESCRIPTION:
The registry collect all the laypeople's performance of 1-minute of chest-compression only CPR registered at the end of a CPR/AED course in which feedback devices were used for at least 1 minute.

All centers which carry out BLS/AED course for laypeople using CPR feedback devices can join to the registry.

All the centers have to declare the duration of the course, the guidelines followed, the participants' anthropometric variables and the feedback device they used for the course and for the test.

The centers must send the performances of all the participants of a course.

ELIGIBILITY:
Inclusion Criteria:

* Layperson
* Participating in a BLS/AED course carried out with feedback devices

Exclusion Criteria:

* Healthcare personnel

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the layperson between 18 and 90 years who participate to a BLS/AED course carried out with the use of feedback devices for at least one minute in one of the centers which joined the registry
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of adequate depth compression | 1 minute
  Percentage of compression performed between 50 and 60 mm for each participant

SECONDARY OUTCOMES:
Mean compression depth | 1 minute
  Mean compression depth for each participant
Percentage of adequate rate compression | 1 minute
  Percentage of compression performed between 100 and 120 per minute for each participant
Compression per minute | 1 minute
  Number of compressions per minute
Percentage of correctly released compression | 1 minute
  Percentage of compressions performed with complete chest recoil
Percentage of correct hand position | 1 minute
  Percentage of compressions performed with hands in the correct position

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (3):
  - Robbio nel Cuore, Robbio, Pavia
  - Policlinico P. Giaccone, Palermo
  - Pavia nel Cuore, Pavia
- Switzerland (2):
  - FormaMed, Cortaillod
  - ES ASUR, Le Mont-sur-Lausanne